CLINICAL TRIAL: NCT06809894
Title: Improvement of the Delirium Management in Adult Patients Hospitalized Through the Use of Non-pharmacological Interventions
Brief Title: Management of Non-pharmacologic Delirium With the Use of a Nursing-led E-health Project: a Randonmized Controlled Trial
Acronym: Delirium
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Collaborators: Hospital d'Igualada (Other)
Responsible Party: Principal Investigator, Laia Fernandez Parra, Registred Nurse (RN) and MSc, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR098/24 (CSA PR35/2023)
Record Dates: First submitted 2025-01-26; First posted 2025-02-05 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Delirium Treatment; Delirium Confusional State; Delirium in Old Age
Keywords: Delirium; SCA; CAM; Older pacient; non-pharmacologic treatment; nurse
MeSH Terms: conditions — Confusion; Delirium | interventions — Educational Status; Nursing Assessment; Vision, Ocular; Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: The study is developed through an experimental cases-control study, developing a quantitative model. A quantitative study is carried out in which the indicators described in the description of the study are studied in order to assess the effectiveness of the implementation of a delirium protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quantitative study for the evaluation of the protocol's effectiveness (Experimental): A quantitative study is carried out in which the indices described in the description of the study are studied in order to assess the effectiveness of the implementation of delirium.
  Interventions: Procedure: Application of an action protocol for the management of delirium through the use of non-pharmacological interventions
- Traditional ways to delirium management (Active Comparator): The use of traditional ways to manage the delirium in hosoitalized older patient, based especially in the use of pharmacological interventions and mechanical patient restraint were compared with the new interventions includes in the new protocol to valorate the effectiveness of the new way to management delirium based in non-pharmacological interventions.
  Interventions: Other: Tradicional management of delirium

INTERVENTIONS:
Procedure: Application of an action protocol for the management of delirium through the use of non-pharmacological interventions — The interventions carried out stand out for being non-pharmacological, this avoiding the use of drugs and polypharmacy in elderly patients, avoiding the appearance of clinical complications derived from the side effects that the use of these substances can lead to in the patient. In addition, it also encourages the education of health professionals and nurses' families or caregivers in the management of delirium.
  Other Names: orientation; mobilitzation; education; feeding assistance; Hypoxemia; Pain; fluid repletion; Therapeutic activities; Nursing Assessment and Intervention Interdisciplinar; Sleep enhancement; Vision and hearing adaptation
  Arms: Quantitative study for the evaluation of the protocol's effectiveness
Other: Tradicional management of delirium — The use of the pharmacological treatment and the mechanical patients restrain were de base of the traditional treatment in deliriums patient in the University hospital of Igualada, because of the less knowledge of the professionals and non-existence protocol of non-pharmacological interventions to management the delirium.
  Other Names: pharmacology; mechanical restrain
  Arms: Traditional ways to delirium management

SUMMARY:
Application of an action protocol focused on the application of non-pharmacological interventions for managing delirium in the process of prevention, diagnosis and treatment, evaluated using an e-health intervention, with a tablet to introduce on it the data about the prevention, diagnostic and treatment process of each recluted patient, in the Igualada Hospital Center, once a day.

DETAILED DESCRIPTION:
1. Generalities Delirium, also known as acute confusional syndrome (ACS), is one of the most common complications in hospitalized patients because its underdiagnosed, increased dependence on basic activities of daily living (ADLs), morbidity and mortality, with nearly 23 deaths per 100 patients diagnosed with delirium. It affects up to 40% of patients over 65 years of age.

   Its occurrence is more frequent in specific hospital settings, such as intensive care units (ICU), emergency departments, or units treating respiratory conditions.

   Several risk factors contribute to the development of delirium, including age (patients over 65 are at higher risk), gender (it is more common in men), polypharmacy, and invasive procedures like bladder catheterization. Patients with urinary tract infections (UTIs) or strictures also face an increased risk.

   In addition, comorbidities like diabetes, stroke, heart failure, or COPD increases the risk of tdeveloping delirium.

   The duration of delirium symptoms can be hours to days, in the 80% of cases, and 20% lasting weeks or even months (4).

   To minimize its impact, it's crucial to focus on proper prevention, early detection, and effective management. A non-pharmacological approach to treatment is key, as reducing medication use can help prevent adverse effects that may worsen the patient's condition.

   Provide adequate training and education for healthcare professionals is essential. To reduce the incidence of delirium in hospitalized patients, a protocol has been developed for its prevention, detection, and treatment through non-pharmacological interventions.
2. Aims General aim To reduce the incidence of delirium through the management of non-pharmacological therapy in the geriatric unit of professionals at the University Hospital of Igualada in the prevention, diagnosis and treatment of hospitalized elderly patients, using a nursing-led e-health intervention.

   2.1. Specific aims To determine whether there are differences in the incidence of delirium with the application of an e-health tablet program, comparing ta control group to and intervention group.
   * To reduce unnecessary pharmacology in patients with delirium of the interventional group comparing to the control group, by promoting the use of non-invasive therapies.
   * To reduce the incidence of delirium in the hospital in the geriatric hospitalization unit.
   * To guarantee an early diagnosis of delirium in hospitalized patients over 80 years of age, with risk criteria, using the CAM scale.
3. Scope of application The application of the protocol is aimed at the University Hospital of Igualada, at the internal medicine units, with the possibility of extrapolating to other units or health centers.

   The protocol is aimed at nurses in the geriatric unit and may receive help from other professionals such as rehabilitation, cleaning, or medical staff in collaborating in the development of the activities.
4. Population and sample The population will include the total number of patients admitted to geriatric unit.

   The patient sample will consist of those who have at least three risk factor for developing delirium, such as age (over 80 years old), gender (male), or benzodiazepines treatment.

   The total sample size will be 65 patients, 32 in the control group and 33 in the intervention group, calculated using the QuestionPro website, based on a population of 77 diagnosed delirium cases in the study units over a 6-month period in 2024 (information provided by the HUI research team). This tool has a margin of error of 5% and a confidence level of 95%.

   The intervention will be carried out by the IP, who is the owner of the development of the e-health application.

   4.1. Inclusion/exclusion criteria Inclusion criteria: Age over 80 years, 3 or more risk factors, admission on geriatric unit in Igualada Hospital Center and social support during the hospital admission.

   Exclusion criteria: Age under 80 years, not presence of risk factors or less than 3, delirium diagnosis in their admission or earlier and foreseeable death on admission not caused by delirium.
5. Data collection and analysis Data collection will be carried out through the completion of the activities about prevention, diagnosis and treatment of delirium through the use of the e-health. The IP and their informatic support will create and app to introduce in a tablet for this purpose.

The data collection will be carried out by the IP once a day, in the morning, during 3 days for each patient of the intervention group.

The data entered into these forms will be automatically transferred into an Excel document with their download in the app. This document will be downloaded by the center's IT team at 3 months after the protocol is implemented, for further analysis.

The Excel document will display the results from each intervention and scale's results, categorized into the following items for further evaluation of the indicators:

* Number of patients at risk of delirium (including those who are subsequently diagnosed and those who are not): This is the number of patients who have risk criteria, without the realization of the CAM scale.
* Number of patients diagnosed with delirium: This is the number of patients with risk criteria, and a positive CAM scale.
* Number of patients with a score of less than 16 on the DRS-R-98 scale: This is the number of patients diagnosed with delirium but with remission of the severity of this clinic, assessed by DRS-R-98.
* Number of days diagnosed with delirium: Of the total number of days hospitalized, how many with delirium.
* Total number of days hospitalized: Total number of days hospitalized.
* Number of patients receiving treatment for delirium: Total number of patients receiving non-pharmacological and pharmacological treatment for delirium.
* Number of patients with drug use for treatment: Of the patients receiving non-pharmacological treatment for delirium, how many need drugs.

Below are the indicators that will be used for the analysis of the data:

INDICATOR 1 Indicator: Rate of patients at risk of developing delirium Zone: Geriatric unit Quality criteria Any patient, on the control or intervention group, presenting symptomatology equivalent to delirium must be assigned this diagnosis.

Definitions: The CAM scale is the reference scale for making the diagnosis of delirium in patients, assessing affirmative answers in 3 or 4 of its items.

Justifications: The diagnosis is made using the CAM scale, assessed once there is a suspicion of the diagnosis, which serves as an element in the diagnosis of the disease. It is recorded using the center's computer program.

Target population: Hospitalized patients over 80 years of age with 3 or more risk factors for the development of delirium.

Formula: Numerator: No. of patients with delirium* 100 / Denominator: Total number of assessed risk patients Type of indicator: Result Data source: Registered in e-health tablet program. Responsible: IP

Periodicity:

* On the appearance of symptoms
* Every 24 hours in the e-healt tablet program, individually for each patient who requires it.
* Quarterly

INDICATOR 2 Indicator: Rate of patients diagnosed with delirium who improve their clinical severity Zone: Geriatric unit Quality criteria: All patients, in the control or intervention group, diagnosed with delirium, must be treated and their symptomatology reduced, assessing the severity of the symptoms.

Definitions: The DRS-R-98 scale assesses the severity of clinical delirium with the evaluation of 7 items, rated from 0 to 4. A higher score indicates more severity, up to 48 points.

Justification: Through DRS-R-98, the severity of the clinical condition is assessed and whether it improves with the application of non-pharmacological therapy. Recorded in the center's computer program, every 24 hours.

Any score equal to or less than 16 will be considered a favorable score, and therefore, a seriousness of the clinic. On the contrary, scores equal to or higher than 17 points, up to a maximum of 48, will indicate a serious severity.

Target population: Hospitalized patients over 80 years old diagnosed with delirium.

Formula: Numerator: No. of patients with a score of less than 16 on the DRS-R-98 scale * 100 / Denominator: No. of patients diagnosed with delirium Type of indicator: Process Data source: Registered on SAVAC program. Responsible: IP

Periodicity:

* Every 24 hours in the e-health tablet program, individually for each patient who requires it.
* Quarterly

INDICATOR 3 Indicator: Rate of drug use in the treatment of delirium Zone: Geriatric unit Quality: All patients, in the control or intervention group, diagnosed with delirium and treated must be able to reduce their hospital stay.

Definitions: Patients diagnosed with delirium tend to have longer hospital stays due to this diagnosis if they are not treated.

Justification: It is assessed on the basis of the number of days spent in hospital, recorded in the patient's clinical history.

Target population: Hospitalized patients over 80 years old diagnosed with delirium.

Formula: Numerator: No. of days with a diagnosis of delirium* 10 / Denominator: Total number of hospitalized days Type of indicator: Result Data source. Clinical history Responsible: IP Periodicity: Quarterly

5. Activities that protocol includes This activities will be included on the e-health tablet program, and for each patient of the intervention group, the IP can select the activities that include in their healthcare during the intervention.

5.1. Prevention

Prevention will be applied to all patients who are admitted to the units where the protocol is applied and present at least 3 risk factor for the development of delirium. As risk factors, they will be considered (2):

* Advanced age (over 80 years old).
* Sex: more common in men.
* Sensory deficits.
* Dehydration and malnutrition.
* Cognitive impairment.
* Comorbidities: hypertension, alcohol abuse, chronic pain, terminal illness, etc.
* Functional disorders.

An other precipitant factors:

* Hypoxia.
* Immobilization.
* Conducting invasive processes.
* Drug abuse.
* Environmental and psychosocial management.
* Fractures or trauma.
* Cardiac surgery.
* Recurrent clinical processes: UTI.

The activities classified with the level of evidence (number) and the degreee of evidence (letter) are:

1. Cognitive Stimulation

   * (1, A) Encourage the patient to say their name, the day of the week, and where they are during daily hygiene, meals, or medication, with the help of nursing staff.
   * (1, A) Ask the patient if they know the reason for their admission to the hospital and explain it to them if they do not understand clearly, but do so without making them feel worried or nervous.
   * (1, A) Ask the patient to share facts about their life, such as whether they have children, siblings, what they enjoy doing, etc., during mealtimes when they are comfortable. This can be done by auxiliary nursing staff.
2. Early Mobilization

   * (1, A) Postural changes by nursing and auxiliary nursing staff.
   * (1, A) Encourage the patient to move around as soon as possible, always considering their capabilities.
   * (1, A) Encourage physiotherapy.
3. Optimal Hydration and Nutrition

   * (1, A) Ensure proper water intake during the patient's breaks to prevent dehydration, and encourage drinking water throughout the day.
   * (1, A) Monitor the amount of food the patient consumes by having the nursing staff check the food trays when they collect them and provide food to those patients who are unable to do so themselves.
4. Maintenance of the Sleep-Wake Cycle

   * (1, A) Illuminate the room by opening the windows during the day, between 8 am and 6 pm in the winter, and between 8 am and 9 pm in the spring and summer, to support the circadian rhythm. This task should be carried out by auxiliary and nursing staff when performing the first vital signs and hygiene routines.
   * (1, A) Close the windows and dim the lights at night, from 6 pm in the winter and 7 pm in the spring/summer.
   * (1, A) Maintain silence during the patient's rest, especially after midnight.
   * (1, A) Minimize invasive techniques and entry into the patient's room at night.
   * Minimize the number of visits to the patient's room by nurses to administer medication and try to administer it at scheduled times.
5. Promotion of Spatial and Temporal Orientation

   * (1, A) Use wall panels in front of the patients' beds, one per room. Ensure they are regularly updated and on time, both by nursing staff and assistants.
   * (1, A) Use up-to-date calendars with large, easy-to-read numbers that show the current date, placed beneath the wall or TV in the rooms.
   * (1, A) Keep the room doors open.
   * (1, A) Offer a radio or television to the patient to stay updated with daily news, which they can use during the day until night, after which it should be turned off for rest time. If a radio is used, it should be provided by the patient's family

5.2. Diagnosis The diagnostic starts when a patient have kind of symptomatology that may trigger delirium.

The nurses cannot assign any type of diagnosis to a patient, but they do have at our disposal tools that facilitate this detection and, together with the medical staff, can determine whether the patient has a diagnosis of delirium.

To make the diagnosis, the Confusional Assessment Method (CAM) and Delirium Rating Scale-Revision-98 (DRS-R-98) will be used to assess the symptomatology and severity of the symptoms.

The following is a summary of what characterizes each scale:

* Confusional Assessment Method (CAM): This is characterized by 5 items that define the assessment at the onset of symptomatology, inattention, disorganized thinking and altered level of consciousness. To confirm the diagnosis of delirium, the patient must have a positive response in domains 1 and 2, as well as a positive response in domains 3 or 4 or both.
* Delirium Rating Scale - Revision -98: This is based on quantifying the severity of delirium by assessing the following domains: cognitive, higher order thinking, circadian cycle, accessory symptoms, and clinical characteristics. These domains have different items included in each of them for their assessment. The score for each item can range from 0 to 3, with a total score of 48. A higher score indicates greater severity of delirium, while a score of 0 indicates that the patient does not suffer from delirium.

These will be completed in the e-heakth program for the IP , where these scales will be included in the patient's registration form.

Once completed, and depending on the results obtained, it will be decided whether the patient is a candidate for a diagnosis of delirium, the respective doctor will be notified, and therefore, specific activities for the treatment of symptomatology will be implemented in the patient's care.

5.3. Treatment's intervention Action on the symptoms will be carried out once the patient has been diagnosed with delirium. The activities to be carried out are similar to those developed in the prevention phase, but more focused on improving the patient's cognitive status.

They will be conducted, once again, bby IP, without leaving aside other professionals such as rehabilitation, physiotherapy or doctors who may collaborate in their development.

The activities classified with the level of evidence (number) and the degreee of evidence (letter) are:

1. Cognitive Stimulation

   • (1, A) Enable relatives to visit the patient to keep their social circle close, at specific times.

   In the case of Covid-19, daily video calls at a set time. Talk to the nursing team and the family to arrange visiting hours or video calls, preferably before bedtime, as this is when the patient is most alert, especially after dinner, to ensure the patient gets a good night's rest.

   • (1, A) Ask the patient to tell us their full name, the day of the week, and where they are.

   This should be done during hygiene routines or when food is served, both by nurses and nursing assistants.
   * (1, A) Management of the sleep-wake cycle. Maintain quiet during the night to support the patient's rest.
   * (1, A) Avoid entering the room during the night as much as possible.
   * (1, A) Open the shutters and let daylight into the room during the day, from 8 am to 6 pm in the late afternoon and winter, and from 8 am to 9pm during spring and summer.
2. Physical Exercises

   • (1, A) Whenever possible, allow the patient to walk around the room before each treatment to prevent hunger or tiredness.

   Encourage physiotherapy.

   • (1, A) Enhance exercise routines. Physical exercises in bed or at the bedside, if standing is not tolerated, such as pulling up the bed, moving the arms, etc.

   Encourage physiotherapy.
3. Orientation Management

   * (1, A) Constantly remind the patient where they are and why.
   * Talk to the patient about where they are and why they are in the hospital during moments of intimacy and trust, such as during hygiene procedures or dressing times, especially by nursing assistants.

Take advantage of moments when injuries are being treated or medication is being administered, especially by nurses.

* (1, A) Always introduce yourself when entering the room and identify yourself as the relevant healthcare staff (nurse, nursing assistant, etc.).
* (1, A) Let the patient know the time and day whenever possible when entering the room.

  d. Music Therapy
* (1, A) Play music that the patient enjoys. Ask about their musical preferences and talk to the family so they can listen to a radio station

5.4. Assessment of symptoms The assessment of symptoms will be carried out by the nursing staff every 48 hours after the diagnosis of delirium until the patient is discharged from the unit.

This will be the last phase of the application of the protocol, assessing the fluctuation of symptomatology and the effectiveness of the activities conducted.

This phase will be completed with the new completion of the DRS-R-98 scale in the program, as soon as the tasks in the infirmary are completed.

The results of the data, as well as the indicators and subsequent evaluation of the impact of the protocol, will be carried out by the hospital supervisor.

ELIGIBILITY:
Inclusion criteria:

* Age over 80 years
* Three risk factor to develop delirium, for example: sex (men), polypharmacy,urinary tract infections (UTIs) or strictures.
* Admission in geriatric unit.
* Have social support

Exclusion criteria:

* Age under 80 years
* Eseeable death on admission not caused by delirium or delirium diagnosis on admission.

Ages: 80 Years to 130 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who develop delirium | Its calculation is carried out during the 3 months of the study, and within each particular case, It is carried out in the morning every day, from admission to discharge of the patient, up to 3 days.
  It is performed on all patients admitted to geriatric unit with 3 or more risk criteria for the development of delirium. Its measurement is carried out in the morning shift using the Confussional Assesment Scale scale. The score is from 0 to 4 points, with a positive diagnosis being one with a score greater than 2. It compares the incidence of the control group and the intervention group.
Rate of patients diagnosed with delirium improving clinical severity | Its calculation is carried out during the three months of the study, and within each particular case, in the morning every day, from the beginning of diagnosis to the improvement of the patient, up to 3 days.
  Every patient with a positive diagnostic and an active treatment. The objective is to avaluate the reduction of the symptoms with the Delirium Rating Scale-R-98 scale, in the morning, comparing control gropu and interventional group . The score is from 0 to 48 points, with a positive diagnosis with severity symptoms in scores greater than 12 points.
Drug use rate for the treatment of delirium | Its calculation is carried out during the 3 months of the study, and within each particular case, in the end of the patient hospitalitzation, up to 3 days.
  Carried out with the recorded on the e-health program and the observation of the clinical history of each patient who have had a positive diagnosis of delirium in their hospitalitzation in the geriatric unit and has recorded the use of drugs, like number of a day and type of drug, for their treatment. Comparation control group and intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Laia Fernandez Parra, Registred Nurse (RN) and MSc, Principal Investigator — Universitat de Lleida; Gloria Tort Nassarre, Registred Nurse (RN), PhD, Study Director — Universitat de Lleida; Aida Bonet Auge, Registred Nurse (RN) and PhD, Study Director — Universitat de Lleida
Locations (1):
- Hospital d'Igualada, Igualada, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data management plan ID 2872, University of Lleida. Only team researchers related to the project will have access to the data.
Supporting Information: Study Protocol
Time Frame: 1 March 2026, start of patient recruitement, it is estimated that it will take approximately 3 months to collect the entire necessary sample.
  The total sample is estimated to be completed in June 2027.
Access Criteria: IP Laia Fernández Parra. Doctoral thesis supervisors, Gloria Tor Nassarre and Aida Bonet Auge. Only data strictly necessary for the project will be accessed. The instructions of the ethics committee are followed.
URL: https://dmp.csuc.cat/plans/2872

REFERENCES:
- [Background] Trzepacz PT, Mittal D, Torres R, Kanary K, Norton J, Jimerson N. Validation of the Delirium Rating Scale-revised-98: comparison with the delirium rating scale and the cognitive test for delirium. J Neuropsychiatry Clin Neurosci. 2001 Spring;13(2):229-42. doi: 10.1176/jnp.13.2.229. PMID 11449030
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Wu YC, Tseng PT, Tu YK, Hsu CY, Liang CS, Yeh TC, Chen TY, Chu CS, Matsuoka YJ, Stubbs B, Carvalho AF, Wada S, Lin PY, Chen YW, Su KP. Association of Delirium Response and Safety of Pharmacological Interventions for the Management and Prevention of Delirium: A Network Meta-analysis. JAMA Psychiatry. 2019 May 1;76(5):526-535. doi: 10.1001/jamapsychiatry.2018.4365. PMID 30810723
- [Background] Ludolph P, Stoffers-Winterling J, Kunzler AM, Rosch R, Geschke K, Vahl CF, Lieb K. Non-Pharmacologic Multicomponent Interventions Preventing Delirium in Hospitalized People. J Am Geriatr Soc. 2020 Aug;68(8):1864-1871. doi: 10.1111/jgs.16565. Epub 2020 Jun 12. PMID 32531089
- [Background] Wilson JE, Mart MF, Cunningham C, Shehabi Y, Girard TD, MacLullich AMJ, Slooter AJC, Ely EW. Delirium. Nat Rev Dis Primers. 2020 Nov 12;6(1):90. doi: 10.1038/s41572-020-00223-4. PMID 33184265
- [Background] Sánchez A, Abdelnour C, Giraldo M, et al. Guia d'abordatge del delirium. Pla de demències de Catalunya. 2022. 1-50.
- [Background] Tobar E, Alvarez E. Delirium in hospitalised older adults. Revista médica clínica Las Condes . 2020;31(1):28-35.
- [Background] Gallardo Navarro M, Martínez Martín M. Delirium in institutionalised elderly: a silent epidemic. Gerokomos . 2023 ;34(1):38-45.
- [Background] Hshieh TT, Inouye SK, Oh ES. Delirium in the Elderly. Clin Geriatr Med. 2020 May;36(2):183-199. doi: 10.1016/j.cger.2019.11.001. PMID 32222295
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32222295/
- See also: Related Info — https://scielo.isciii.es/pdf/geroko/v34n1/1134-928X-geroko-34-01-38.pdf
- See also: Related Info — https://www.nature.com/articles/s41572-020-00223-4.pdf